CLINICAL TRIAL: NCT06553534
Title: Situation Awareness Incorporating Multidisciplinary Teams Reduce Arrests In the Pediatric ICU in the Pediatric Resuscitation Quality Collaborative
Brief Title: Situation Awareness Incorporating Multidisciplinary Teams Reduce Arrests In the Pediatric ICU
Acronym: SAMURAI PICU
Status: Active, not recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Children's Hospital Medical Center, Cincinnati (Other)
Collaborators: Children's Hospital of Philadelphia (Other); Agency for Healthcare Research and Quality (AHRQ) (U.S. Federal Agency)
Responsible Party: Sponsor
Allocation: Randomized | Model: Crossover | Masking: None | Purpose: Prevention
Other Study IDs: SAMURAI_23-021338; 1R18HS029630-01 (AHRQ)
Record Dates: First submitted 2024-08-12; First posted 2024-08-14 (Actual); Last update posted 2024-08-16 (Actual); Status verified 2024-08

CONDITIONS: In-hospital Cardiac Arrest; Cardiopulmonary Resuscitation
Keywords: situational awareness; Cardiac Arrest; Cardiopulmonary Resuscitation
MeSH Terms: conditions — Heart Arrest

STUDY DESIGN:
Intervention Model Description: Adaptive Hybrid Stepped-wedge
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (5):
- Site A (Experimental): Site A will begin a transition period of no more than 6 months (while continuing to collect baseline data). During the transition period, the local study team will receive education about the intervention and help tailor the tools and materials to fit their institutional needs. Upon completion of the transition period, Site A will immediately begin the intervention period. They will then remain in the intervention period (using the SAMURAI Bundle) for the remaining study period.
  Interventions: Other: SAMURAI PICU Bundle
- Site B (Experimental): Site B will begin a control period of approximately 6 months, during which they will continue to collect data while operating under their institutional standards (No SAMURAI Intervention). At the end of the control period, they will start a transition period of up to 6 months, during which time they will receive education and adapt the tools and materials to fit their institutional needs. At the conclusion of the transition period, they will begin implementing the study intervention (usage of the SAMURAI bundle) for the remaining study period
  Interventions: Other: SAMURAI PICU Bundle
- Site C (Experimental): Site C will begin a control period of approximately 1 year, during which they will continue to collect data while operating under their institutional standards (No SAMURAI Intervention). At the end of the control period, they will start a transition period of up to 6 months, during which time they will receive education and adapt the tools and materials to fit their institutional needs. At the conclusion of the transition period, they will begin implementing the study intervention (usage of the SAMURAI bundle) for the remaining study period.
  Interventions: Other: SAMURAI PICU Bundle
- Site D (Experimental): Site D will begin a control period of approximately 1.5 years, during which they will continue to collect data while operating under their institutional standards (No SAMURAI Intervention). At the end of the control period, they will start a transition period of up to 6 months, during which time they will receive education and adapt the tools and materials to fit their institutional needs. At the conclusion of the transition period, they will begin implementing the study intervention (usage of the SAMURAI bundle) for the remaining study period.
  Interventions: Other: SAMURAI PICU Bundle
- Site E (No Intervention): Site E will serve as our control group for the study period, operating according to their institutional standard of care (No intervention) while continuing to collect data.

INTERVENTIONS:
Other: SAMURAI PICU Bundle — The proposed multifaceted SAMURAI PICU Bundle is an intervention with the following core elements: 1) PICU Warning Tool: an automated clinical decision support (CDS) tool to provide a non-interruptive interprofessional predictive alert, 2) twice daily safety huddles with unit leadership, and 3) bedside assessment including the care team and patient's family to complete and display a bedside mitigation plan to prevent deterioration. This intervention combines the automated accurate prediction of the PICU Warning Tool with the use of provider intuition or a "gut feeling" from huddles to improve decision making at the bedside. Peripheral elements and possible adaptations will be suggested during Aim 1 and additional peripheral elements may be added by local sites after discussion with the PI through a user-centered design approach.
  Other Names: SAMURAI Bundle
  Arms: Site A; Site B; Site C; Site D

SUMMARY:
The goal of this pragmatic prospective Type 1 Hybrid Implementation-Effectiveness Trial study is to learn if The Situation Awareness Incorporating Multidisciplinary Teams Reduce Arrests In (SAMURAI) the PICU Bundle can reduce PICU CPR events. The SAMURAI PICU Bundle includes an automated PICU warning tool, twice daily huddles and mitigation plans. The main questions it aims to answer are:

Is the adapted bundle will be acceptable, feasible, and appropriate to stakeholders prior to implementation?

Will there be at least a 30% relative reduction in PICU CPR events following successful implementation of the bundle?

Each site will:

Adapt and implement SAMURAI PICU Bundle which includes an automated PICU warning tool, twice daily huddles and mitigation plans

DETAILED DESCRIPTION:
As nearly 95% of pediatric IHCAs occur in PICUs, we developed an interventional cardiac arrest prevention bundle targeted to PICU healthcare providers. In a previous single center trial, the use of the SAMURAI PICU bundle improved early identification of high-risk patients, increased shared situation awareness, and supported risk mitigation plans, leading to a >50% decrease in IHCA events requiring cardiopulmonary resuscitation (CPR). Early identification occurs via the PICU Warning Tool, an automated, electronic medical record clinical decision support tool that provides a non-interruptive notification to care providers of high-risk patients. This prediction tool prompts a bedside huddle to ensure shared situation awareness and development of a mitigation plan. This novel approach of emphasizing shared situation awareness through automated clinical decision support and mitigation of risk has demonstrated reduction in CPR events and mortality within the PICU clinical environment.

This study employs a user-centered design model to adapt, implement, and assess the feasibility and effectiveness of SAMURAI PICU at other pediatric institutions. The hypothesis is that identification of PICU patients at high risk for IHCA through the use of the PICU Warning Tool and integration of this high-risk status in daily safety huddles will lead to improved shared situation awareness and subsequent reduction in CPR events at participating institutions. This approach will utilize a five-center pragmatic prospective Hybrid Type 1 effectiveness-implementation study leveraging the existing infrastructure of Pediatric Resuscitation Quality Collaborative (pediRES-Q).

ELIGIBILITY:
Inclusion Criteria:

* All patients admitted to the five PICUs in pediRES-Q during the study period

Exclusion Criteria:

* None

Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Enrollment: 5 (Actual)
Dates: Start 2024-01-01 (Actual); Primary Completion 2029-01 (Estimated); Study Completion 2029-01 (Estimated)

PRIMARY OUTCOMES:
Effectiveness - CPR Event Rate | 2 years and 4 years
  The primary outcome is CPR Event Rate per 1000 Patient Days. CPR Events will be defined per Utstein Criteria.

CONTACTS AND LOCATIONS:
Overall Officials: Maya L Dewan, MD, MPH, Principal Investigator — Children's Hospital Medical Center, Cincinnati
Locations (5):
- United States (5):
  - Comer Children's Hospital, Chicago, Illinois
  - Akron Children's Hospital, Akron, Ohio
  - MUSC Shawn Jenkins Children's Hospital, Charleston, South Carolina
  - Children's Hospital of Richmond, Richmond, Virginia
  - Seattle Children's, Seattle, Washington

REFERENCES:
- [Background] Molloy MJ, Zackoff M, Gifford A, Hagedorn P, Tegtmeyer K, Britto MT, Dewan M. Usability Testing of Situation Awareness Clinical Decision Support in the Intensive Care Unit. Appl Clin Inform. 2024 Mar;15(2):327-334. doi: 10.1055/a-2272-6184. Epub 2024 Feb 20. PMID 38378044
- [Background] Gifford A, Butcher B, Chima RS, Moore L, Brady PW, Zackoff MW, Dewan M. Use of design thinking and human factors approach to improve situation awareness in the pediatric intensive care unit. J Hosp Med. 2023 Nov;18(11):978-985. doi: 10.1002/jhm.13216. Epub 2023 Oct 4. PMID 37792360
- [Background] Dewan M, Soberano B, Sosa T, Zackoff M, Hagedorn P, Brady PW, Chima RS, Stalets EL, Moore L, Britto M, Sutton RM, Nadkarni V, Tegtmeyer K, Wolfe H. Assessment of a Situation Awareness Quality Improvement Intervention to Reduce Cardiac Arrests in the PICU. Pediatr Crit Care Med. 2022 Jan 1;23(1):4-12. doi: 10.1097/PCC.0000000000002816. PMID 34417417
- [Background] Soberano BT, Brady P, Yunger T, Jones R, Stoneman E, Sosa T, Stalets EL, Zackoff M, Chima R, Tegtmeyer K, Dewan M. The Effects of Care Team Roles on Situation Awareness in the Pediatric Intensive Care Unit: A Prospective Cross-Sectional Study. J Hosp Med. 2020 Oct;15(10):594-597. doi: 10.12788/jhm.3449. PMID 32853138